CLINICAL TRIAL: NCT06709651
Title: Prospective Evaluation of the Breast Microbiome and Tumor Microenvironment-related Biomarkers of Response to Neoadjuvant Systemic Therapy in Triple Negative Breast Cancer
Brief Title: Microbiome Immunotherapy Neoadjuvant Assessment
Acronym: MINA
Status: Recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 23120
Record Dates: First submitted 2024-11-01; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast tissue biopsy, blood and stool samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Predictive biomarkers of response to combination chemotherapy and immune-checkpoint inhibitors are urgently needed to help tailor treatment recommendations for patients with early-stage TNBC. Tumour-associated microbiota in primary breast tumours represent promising and novel candidate biomarkers modulators of the efficacy of therapies for patients with TNBC. It has been shown that microbes colonizing breast tumours can modulate the efficacy of commonly used drugs and that the microbiome of breast tissue biopsies could represent a new biomarker. Data on the microbiome of patients with cancer indicate the potential for a new class of bacteria-based oncological biomarkers, for exploitation in precision oncology.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial in accordance with national/local guidelines.
2. Be a male or female subject 18 years of age on day of signing informed consent.
3. Histologically proven infiltrating carcinoma of the breast on core needle biopsy that is:

   HER2 negative in primary tumour pre-treatment by local pathology assessed according current ASCO/CAP guidelines: In situ hybridization non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell), OR Immunohistochemistry (IHC) 0 or IHC 1+.

   ER and PR negative in primary tumour pre-treatment defined as < 10% of cells expressing hormonal receptors via IHC analysis by local laboratory assessment.
4. Unresected, untreated breast cancer planned to undergo neoadjuvant systemic therapy, that meets one of the following clinical stages (see Appendix A):

   o T2, T3, or T4a-d lesion, any N, M0
5. Be willing to undergo mandatory research biopsy procedure at baseline (up to 4 core samples may be taken from this procedure).

Exclusion Criteria:

1. Patients who are pregnant or breast-feeding
2. Current use of any investigational agents
3. History or current evidence of any condition, therapy, lab abnormality or other circumstance that in the opinion of the investigator might expose the subject to risk by participating in the trial, confound the results of the trial, or interfere with the subject's participation for the full duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Cork University Hospital that meet inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the breast cancer microbiome pre- and post-therapy, in patients with early stage TNBC undergoing neoadjuvant systemic therapy | Through study completion, an average of 1 year
  Microbiome evaluation with metagenomic sequencing to assess changes in the relative abundance of microbial taxa (measured as percentage abundance per microbial species and changes in percentage abundance between baseline and post-therapy timepoints)

SECONDARY OUTCOMES:
To examine the relationship between the local breast cancer microbiome in early-stage triple negative breast cancer and pathologic complete response | Through study completion, an average of 1 year
  Correlation between breast microbiome composition (measured as percent abundance of microbial taxa derived from metagenomic sequencing) and pathologic complete response rate (pCR)
To examine the relationship between the local breast cancer microbiome in early-stage triple negative breast cancer and event-free survival | Through study completion, an average of 1 year
  Correlation between breast microbiome composition (measured as percent abundance of microbial taxa derived from metagenomic sequencing) and event free survival (EFS)
To examine the relationship between the local breast cancer microbiome in early-stage triple negative breast cancer and overall survival | Through study completion, an average of 1 year
  Correlation between breast microbiome composition (measured as percent abundance of microbial taxa derived from metagenomic sequencing) and overall survival (OS)
To determine the relationship between the breast cancer microbiome and tumor infiltrating leukocytes (TILs) | Through study completion, an average of 1 year
  Correlation between breast microbiome composition (measured as percent abundance of microbial taxa derived from metagenomic sequencing) and TILS (<50% versus ≥50%)
To determine the relationship between the breast cancer microbiome and programmed death ligand -1 (PDL-1) | Through study completion, an average of 1 year
  Correlation between breast microbiome composition (measured as percent abundance of microbial taxa derived from metagenomic sequencing) and , PDL1 (positive defined as CPS ≥ 1 by PD-L1 IHC 22C3 assay versus negative)
To evaluate the gut microbiome pre- and post-therapy, in patients with early stage TNBC undergoing neoadjuvant systemic therapy | Through study completion, an average of 1 year
  Change in the gut microbiome composition (measured as percent abundance of microbial taxa derived from metagenomic sequencing) between pre- and post-therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Undecided